CLINICAL TRIAL: NCT06543485
Title: Results of Intramedullary Headless Screw Fixation for Metacarpal Fractures in Adults.
Brief Title: Headless Screw Fixation for Metacarpal Fractures in Adults.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohannad Bahaa Al-Sayyd, Resident of Orthopaedics and Traumatology, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-24-07-13MS
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Metacarpal Fractures in Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adults with metacarpal fractures (Experimental): intramedullary screw fixation of metacarpal fractures
  Interventions: Procedure: intramedullary screw fixation of metacarpal fractures

INTERVENTIONS:
Procedure: intramedullary screw fixation of metacarpal fractures — intramedullary screw fixation of metacarpal fractures through limited open approach

SUMMARY:
The goal of this study is to evaluate results of intramedullary screw fixation of metacarpal fractures while summarizing the pearls and pitfalls to maximize successful surgical outcomes in adults, Metacarpal fractures are third most common upper extremity fractures, Intramedullary screw Fixation is a fixation option that offers rigid stability, early active range of motion, and simplicity of insertion,

ELIGIBILITY:
Inclusion Criteria:

* Adult patients.
* Metacarpal shaft fractures.
* Simple fractures.
* Recent fractures within 1-2 weeks.
* Isolated metacarpal fractures.

Exclusion Criteria:

* Pediatric fractures with open physis.
* Head-splitting fractures and Metacarpal basal fractures.
* Compound fracture increasing risk of infection.
* medical illness or mental disorders affecting the follow-up examination.
* Association with other fractures fixed by methods that limit early range of motion.
* pathologic fractures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
early active range of motion | 3 days-12 weeks after surgery
  QuickDASH score ( Disabilities of the Arm, Shoulder and Hand questionnaire )

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Select A State Or Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nakashian MN, Pointer L, Owens BD, Wolf JM. Incidence of metacarpal fractures in the US population. Hand (N Y). 2012 Dec;7(4):426-30. doi: 10.1007/s11552-012-9442-0. PMID 24294164
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787
- [Background] Karl JW, Olson PR, Rosenwasser MP. The Epidemiology of Upper Extremity Fractures in the United States, 2009. J Orthop Trauma. 2015 Aug;29(8):e242-4. doi: 10.1097/BOT.0000000000000312. PMID 25714441
- [Background] Chung KC, Spilson SV. The frequency and epidemiology of hand and forearm fractures in the United States. J Hand Surg Am. 2001 Sep;26(5):908-15. doi: 10.1053/jhsu.2001.26322. PMID 11561245
- [Background] Page SM, Stern PJ. Complications and range of motion following plate fixation of metacarpal and phalangeal fractures. J Hand Surg Am. 1998 Sep;23(5):827-32. doi: 10.1016/S0363-5023(98)80157-3. PMID 9763256
- [Background] Robinson LP, Gaspar MP, Strohl AB, Teplitsky SL, Gandhi SD, Kane PM, Osterman AL. Dorsal versus lateral plate fixation of finger proximal phalangeal fractures: a retrospective study. Arch Orthop Trauma Surg. 2017 Apr;137(4):567-572. doi: 10.1007/s00402-017-2650-x. Epub 2017 Feb 24. PMID 28236187
- [Background] Siddiqui AA, Kumar J, Jamil M, Adeel M, Kaimkhani GM. Fixation of Metacarpal Fractures Using Intramedullary Headless Compression Screws: A Tertiary Care Institution Experience. Cureus. 2019 Apr 16;11(4):e4466. doi: 10.7759/cureus.4466. PMID 31249744
- [Background] Botte MJ, Davis JL, Rose BA, von Schroeder HP, Gellman H, Zinberg EM, Abrams RA. Complications of smooth pin fixation of fractures and dislocations in the hand and wrist. Clin Orthop Relat Res. 1992 Mar;(276):194-201. PMID 1537152
- [Background] Stahl S, Schwartz O. Complications of K-wire fixation of fractures and dislocations in the hand and wrist. Arch Orthop Trauma Surg. 2001 Oct;121(9):527-30. doi: 10.1007/s004020100279. PMID 11599756
- [Background] Eberlin KR, Babushkina A, Neira JR, Mudgal CS. Outcomes of closed reduction and periarticular pinning of base and shaft fractures of the proximal phalanx. J Hand Surg Am. 2014 Aug;39(8):1524-8. doi: 10.1016/j.jhsa.2014.05.008. Epub 2014 Jul 2. PMID 24996674
- [Background] Hoang D, Vu CL, Jackson M, Huang JI. An Anatomical Study of Metacarpal Morphology Utilizing CT Scans: Evaluating Parameters for Antegrade Intramedullary Compression Screw Fixation of Metacarpal Fractures. J Hand Surg Am. 2021 Feb;46(2):149.e1-149.e8. doi: 10.1016/j.jhsa.2020.08.007. Epub 2020 Oct 19. PMID 33092908